CLINICAL TRIAL: NCT03946241
Title: Physical Activity in Schools After the Reform
Acronym: PHASAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry); University of Cambridge (Other)
Responsible Party: Principal Investigator, Anders Groentved, Associate professor, University of Southern Denmark
Other Study IDs: 72682; 115606 (Other Grant/Funding Number: TrygFonden)
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Physical Activity; Overweight; Physical Inactivity
Keywords: School children; Physical Activity; Accelerometry; Body mass index; Implementation; Policy
MeSH Terms: conditions — Motor Activity; Overweight; Sedentary Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-reform study populations: Children from 1st to 9th grade (n ~ 2,600) from four different school-based studies collecting objective physical activity data. The four studies are 1) The European Youth Heart Study (EYHS) conducted in 1997-98, 2003-04 and 2009-10, 2) When Cities Move Children (WCMC) conducted in 2010 and 2012, 3) Childhood Health, Activity, and Motor Performance School Study Denmark (CHAMPS-DK) conducted in 2009, 2010 and 2012, and 4) School site, Play Spot, Active transport, Club fitness and Environment (SPACE) conducted in 2010 and 2012. A total of 44 schools where included in the studies.
- Post-reform study population: Children from 1st to 9th grade in 2017-18 from the same schools as included in the pre-reform research studies (n ~ 2,600). Two of the pre-reform research studies (CHAMPS-DK and SPACE) introduced PA promoting initiatives as part of the study. To minimize any influence from participation in these interventions we chose only to include and recruit participants from control schools from these studies. A total of 36 schools where invited and 31 subsequently accepted to participate. Parents and teachers of the children were included as well.

SUMMARY:
In 2014 the Danish Government introduced a wide-ranging school reform that applies to all public schools in Denmark. In a physical activity promotion perspective, a distinctive feature of the school reform is that it has become mandatory to integrate an average of 45 minutes of daily physical activity in the regular school day. The overarching objective of the PHASAR study is to evaluate the implementation of this ambitious policy-driven physical activity promotion initiative and its potential effect on physical activity and overweight.

The PHASAR study provides a rare opportunity to evaluate the effectiveness of a nation-wide policy-driven school-based physical activity promotion initiative.

DETAILED DESCRIPTION:
In 2014 the Danish Government introduced a wide-ranging school reform that applies to all public schools in Denmark. The reform involved changes in several aspects of the school structure and content. In a physical activity promotion perspective, a distinctive feature of the school reform is that it has become mandatory to integrate an average of 45 minutes of daily physical activity during the regular school day. The overarching objective of the PHASAR study is to evaluate the implementation of this ambitious policy-driven physical activity promotion initiative and the possible effect on children's level of physical activity and overweight. Moreover, by applying improved accelerometry technology, the study aims to provide a detailed characterization of physical activity during the children's entire day including the school day.

The evaluation is divided into a quantitative effect evaluation and a combined quantitative and qualitative process evaluation. A total of 31 schools were enrolled and 2,683 pairs of accelerometers were handed out to school-aged children from 1st to 9th grade in the PHASAR study during the 2017/18 school year. The objectively measured physical activity data will be compared to repeated cross-sectional data collected in four historical school-based studies from 1998-2012. Body mass index data from 2012-2018 will be collected from The Child Database, which includes repeated cross-sectional assessments on approximately 100,000 children annually. In the absence of a control group, interrupted time-series analysis will be used to evaluate pre- and post-reform physical activity and body mass index levels and trends. A characterization of the school environment relevant for physical activity promotion on a political, environmental, organizational and individual level, as well as school implementation processes will be conducted to evaluate the implementation process. Data will be collected using interviews, surveys, document analyses and observations.

The PHASAR study provides a rare opportunity to evaluate the effectiveness of a nation-wide policy-driven school-based physical activity promotion initiative. The use of objectively measured pre- and post-reform physical activity and body mass index data combined with a characterization of the school implementation processes regarding the promotion of physical activity will provide a comprehensive source of information needed to evaluate the school reform.

ELIGIBILITY:
Inclusion criteria:

Pre-reform study population:

- School children who been included in one of the four pre-reform studies.

Post-reform study population:

- Children attended one of the public schools and age groups that had already been included in one of the four pre-reform studies.

Exclusion criteria:

- School children that suffers from physical disabilities or injuries preventing physical activity.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pre-reform studies:
  School children in 1st to 9th grade (ages between 6 and 17 years). The participating children's parents or legal guardians.
  Post-reform studies:
  School children in 1st to 9th grade (ages between 6 and 17 years). The participating children's parents or legal guardians. Teachers, pedagogues, and headmasters from the same schools.
Sampling Method: Non-Probability Sample
Enrollment: 5200 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in levels of school time physical activity, reported as time spent moving, in a representative sample of school children before and after the school reform. | Pre-reform data have been collected between 1998 and 2012. Post-reform data have been collected during the school year 2017 to 2018.
  Objectively measured physical activity data are obtained via accelerometers mounted on the hip of the school children for a representative number of consecutive days. The school children's time spent moving will be longitudinally analysed on the school level (not class or individual level).

SECONDARY OUTCOMES:
Change in school children's BMI from the majority of all Danish public schools before, during, and after implementing the school reform. | National BMI data have been obtained annually from 2011 and onwards. Thus, data from 2011 till 2018 will be utilized for this outcome.
  Height and weight are obtained from the Child Database (Børnedatabasen), which is based on data from the mandatory examinations in schools by school nurses on three occasions during children's years in public school. The first measurement is conducted at the age of 6 to 7 years of age (in case of several measurements, the first was registered). The second measurement is conducted when children were between 9 and 13 years old (in case of several measurements, the measurement closest to the age of 11 was registered). The third measurement is conducted when children were 14 or 15 years old (in case of several measurements, the last was registered).
Changes in BMI among school children before and after implementing the school reform. | Data will be obtained from the pre-reform research studies in the years leading up to the school reform and the data collected during the school years 2017/18 and 2018/19.
  School levels of changes in BMI will be compared in the pre- and post-reform study populations and analysed according to school levels of physical activity (child time spent moving).
Changes in waist-to-height ratio among school children before and after implementing the school reform. | Data will be obtained from the pre-reform research studies in the years leading up to the school reform and the data collected during the school years 2017/18 and 2018/19.
  School levels of changes in waist-to-height ratio will be compared in the pre- and post-reform study populations (were available) and analysed according to school levels of physical activity (child time spent moving).
Change in time spent in moderate to vigorous physical activity in school children during school time, leisure time and total time from before till after the school reform. | Data will be obtained from the pre-reform research studies in the years leading up to the school reform and the data collected during the school years 2017/18 and 2018/19.
  In order to investigate the effect of the school reform on health-related physical activity, change in time spent in moderate to vigorous physical activity (assessed by hip worn accelerometer) for school children before and after the school reform will the analysed.
The total amount of physical activity in school children during school time, leisure time and total time before and after the school reform. | Data will be obtained from the pre-reform research studies in the years leading up to the school reform and the data collected during the school years 2017/18 and 2018/19.
  The total amount of physical activity in school children during school time, leisure time and total time assessed using hip worn accelerometer will be reported as counts per minute for school children before and after the school reform.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grøntved, PhD, Principal Investigator — University of Southern Denmark; Jens Troelsen, Professor, Principal Investigator — University of Southern Denmark
Locations (1):
- Department of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD will be anonymised and handed over to the Danish National Archives. From there researchers can request the database for additional or new analyses.
Supporting Information: Study Protocol, SAP
Time Frame: The data are expected to be available latest on the 1st of august 2027. It is likely that it will be available from approximately 2021. After data has been handed over, there is no expiry of availability.
Access Criteria: For the first 20 years after the data has been handed over to the Danish National Archives the inquirer can get access to the data if the PI of the project accepts the inquiry. After this, there is no restrictions on availability.
URL: http://dda.dk/simple-search

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03946241/SAP_001.pdf